CLINICAL TRIAL: NCT03860818
Title: Improving Transplant Medication Safety Through a Technology and Pharmacist (ISTEP) Intervention in Veterans
Brief Title: Improving Transplant Medication Safety Through A Technology and Pharmacist Intervention
Acronym: ISTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 15-359
Record Dates: First submitted 2019-02-28; First posted 2019-03-04 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-05

CONDITIONS: Transplant
Keywords: medication safety

STUDY DESIGN:
Intervention Model Description: Prospective, cluster-randomized controlled clinical trial at 10 sites, randomizing 5 sites to standard clinical care and 5 to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (No Intervention): Usual Care
- Intervention Arm (Experimental): Technology-enabled pharmacist intervention
  Interventions: Other: Health services delivery

INTERVENTIONS:
Other: Health services delivery — Technology-enabled pharmacist intervention
  Arms: Intervention Arm

SUMMARY:
Medication safety issues in Veteran organ transplant recipients, including side effects and errors, are a major issue leading to graft failure and death. The causes of these events are complicated and involve fragmented care, communication breakdowns between the Veterans, providers and the different health care systems. This grant proposal seeks to improve medication safety within these high-risk Veterans, using two innovative components; the application of technology to leverage the massive amount of data contained within the electronic medical record in identifying Veterans with potential medication safety issues, coupled with a pharmacist-led intervention to improve the management and coordination of immunosuppression therapy. The completion of this prospective, multicenter, cluster randomized controlled clinical trial will provide evidence that these interventions can improve medication safety, clinical outcomes and costs and will be used to justify the dissemination of these interventions to all VAs caring for Veteran transplant recipients across the U.S.

DETAILED DESCRIPTION:
Anticipated Impacts on Veterans Health Care: The first three essential strategies listed within the VA's Blueprint for Excellence encompass plans to improve care to vulnerable Veterans, deliver high quality care through achieving the "Triple Aim" and leverage the use of technology to improve the efficiency of care delivery. The intervention this grant proposes focuses on improving medication safety and care coordination within a high risk vulnerable Veteran population, leverages the use of informatics and analytics to support this intervention, and aims to demonstrate improved care at reduced costs through the pharmacist intervention; thus, perfectly aligning with these three essential components of the Blueprint. The overarching goal of this study is to develop a feasibly deployable, technology-enabled intervention that will demonstrate substantial improvements in immunosuppressant medication safety, clinical outcomes and health care costs in Veteran organ transplant recipients; demonstrating this through a randomized controlled trial will provide sufficient evidence to further develop a VA-specific pharmacist learning collaborative aimed at improving care and reducing costs for Veteran organ transplant recipients across the entire VA system.

Background: Organ transplant is the gold-standard treatment for patients with end organ diseases of the kidney, liver, heart and lungs, as it substantially improves survival and quality of life. Over the past 20 years, the use of contemporary immunosuppression has reduced the risk of acute rejection rates by upwards of 80%; yet long-term allograft survival remains suboptimal. Studies have demonstrated that causes of late graft loss is predominantly driven by immunosuppression adverse events and late allograft rejection episodes from medication errors and non-adherence, which encompass issues directly related to medication safety. The investigators' research demonstrates that medication errors occur in nearly two-thirds of transplant recipients, leading to hospitalization in 1 in 8 recipients. Recipients that develop significant medication errors are at considerably higher risk of graft loss, leading to higher costs and mortality. Thus, in order to improve medication safety and long-term outcomes in transplant recipients, enhancements in immunosuppressant therapy management is needed.

Objectives: The central hypothesis for the ISTEP study (Improving Transplant Medication Safety through a TEchnology and Pharmacist Intervention) is that pharmacist-led immunosuppressant therapy management, facilitated through the use of innovative technology, will significantly improve immunosuppressant safety and clinical outcomes in Veteran transplant recipients.

Methods: This is a 24-month, prospective, cluster-randomized controlled clinical trial at 10 sites, randomizing 5 sites to standard clinical care and 5 to standard care and the technology-enabled pharmacist intervention. The technology component of this intervention consists of the use of an expanded dashboard system that has already demonstrated effectiveness in improving immunosuppression monitoring. The dashboard performs population-level surveillance of transplant recipients and identifies those with potential drug-related problems, including non-adherence, drug interactions, missing and worrisome trends in labs; then providing a real-time alert to the pharmacist, who will determine its relevance and intervene in an appropriate protocol-guided manner. Effectiveness will be determined by comparing the rates of hospitalizations and ER visits between groups, while adjusting for baseline patient, provider and facility characteristics. Secondary measures include comparing healthcare costs and determining dashboard functionality, dashboard actionability and pharmacist intervention types and acceptance rates. The investigators will also assess the overall incidence and severity of drug-related problems and graft and patient survival rates and compare these between the intervention and control sites.

ELIGIBILITY:
Inclusion Criteria:

* Veteran organ transplant recipients will be identified using International Classification of Diseases (ICD) 9/10 codes from the VA electronic health record (CPRS).
* Patients must have an active code stating they are a recipient of an organ transplant.
* The following codes will be utilized - ICD-9 codes:

  * V42.0
  * V42.1
  * V42.6
  * V42.7
  * V42.83
  * V42.84
  * 996.81
  * 996.82
  * 996.83
  * 996.84
  * 996.86
  * 52.80

OR

* oICD-10 codes:

  * C80.2
  * T86.1
  * T86.10
  * T86.11
  * T86.12
  * T86.13
  * T86.19
  * T86.2
  * T86.20
  * T86.21
  * T86.22
  * T86.23
  * T86.290
  * T86.298
  * T86.3
  * T86.30
  * T86.31
  * T86.32
  * T86.33
  * T86.39
  * T86.4
  * T86.40
  * T86.41
  * T86.42
  * T86.43
  * T86.49
  * T86.810
  * T86.811
  * T86.812
  * T86.818
  * T86.819
  * T86.9
  * Z48.2
  * Z48.21
  * Z48.22
  * Z48.23
  * Z48.24
  * Z48.280
  * Z48.288
  * Z48.298
  * Z94.0
  * Z94.1
  * Z94.2
  * Z94.3
  * Z94.4
  * Z94.83

AND

* Actively receiving at least one anti-rejection medication dispensed by the VA site.
* These medications include:

  * tacrolimus
  * cyclosporine
  * azathioprine
  * mycophenolate
  * sirolimus
  * everolimus
  * belatacept

Exclusion Criteria:

* There are no exclusion criteria for patients in this study as recruitment is at the level of the VA site.
* All veterans meeting inclusion criteria will be monitored by the dashboard system and will be included in the outcomes assessment.
* Patients may enter or exit the study in a rolling manner, which will be accounted for during analyses.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2196 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Taber, PharmD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Taber DJ, Ward R, Axon RN, Walker RJ, Egede LE, Gebregziabher M. The Impact of Dual Health Care System Use for Obtaining Prescription Medications on Nonadherence in Veterans With Type 2 Diabetes. Ann Pharmacother. 2019 Jul;53(7):675-682. doi: 10.1177/1060028019828681. Epub 2019 Feb 6. PMID 30724092
- [Result] Taber DJ, Ward RC, Buchanan CH, Axon RN, Milfred-LaForest S, Rife K, Felkner R, Cooney D, Super N, McClelland S, McKenna D, Santa E, Gebregziabher M. Results of a multicenter cluster-randomized controlled clinical trial testing the effectiveness of a bioinformatics-enabled pharmacist intervention in transplant recipients. Am J Transplant. 2023 Dec;23(12):1939-1948. doi: 10.1016/j.ajt.2023.08.004. Epub 2023 Aug 9. PMID 37562577
- [Derived] Hall CL, Fominaya CE, Gebregziabher M, Milfred-LaForest SK, Rife KM, Taber DJ. Improving Transplant Medication Safety Through a Technology and Pharmacist Intervention (ISTEP): Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2019 Oct 1;8(10):e13821. doi: 10.2196/13821. PMID 31573933

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Arm: The control arm received usual care. Usual care for veteran organ transplant recipients across the 10 study sites is not standardized but generally includes the following: at most sites, nurse coordinators and/or midlevel practitioners are responsible for general transplant patient oversight, including ensuring laboratory assessments are scheduled/reviewed and medication regimens are accurate and up to date. However, large patient numbers and workload constraints preclude these health care professionals from prospective detailed daily monitoring of patients. Within usual follow-up care, pharmacists do not conduct routine daily surveillance of all transplant patients.
- Intervention Arm: Technology-enabled pharmacist intervention
  Health services delivery: Technology-enabled pharmacist intervention.
  The intervention consists of increased review of patients by a pharmacist and increased scrutiny of patients' medication regimens and laboratory values using a dashboard surveillance system.
Period: Overall Study
Arm/Group | Control Arm | Intervention Arm
Started | 896 | 1300
Completed | 720 | 1060
Not Completed | 176 | 240
Not completed — Death | 144 | 195
Not completed — Graft Loss | 32 | 45

BASELINE CHARACTERISTICS:
Groups:
- Control Arm: Usual Care. The control arm received usual care. Usual care for veteran organ transplant recipients across the 10 study sites is not standardized but generally includes the following: at most sites, nurse coordinators and/or midlevel practitioners are responsible for general transplant patient oversight, including ensuring laboratory assessments are scheduled/reviewed and medication regimens are accurate and up to date. However, large patient numbers and workload constraints preclude these health care professionals from prospective detailed daily monitoring of patients. Within usual follow-up care, pharmacists do not conduct routine daily surveillance of all transplant patients.
- Intervention Arm: Technology-enabled pharmacist intervention
  Health services delivery: Technology-enabled pharmacist intervention
  The intervention consists of increased review of patients by a pharmacist and increased scrutiny of patients' medication regimens and laboratory values using a dashboard surveillance system.
- Total: Total of all reporting groups
Arm/Group | Control Arm | Intervention Arm | Total
Number analyzed (Participants) | 896 | 1300 | 2196
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67 [60 to 71] | 66 [60 to 71] | 66 [60 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 57 | 98
  Male | 855 | 1243 | 2098
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic White | 608 | 834 | 1442
  Race/Ethnicity: Hispanic | 39 | 47 | 86
  Race/Ethnicity: Non-Hispanic Black | 206 | 386 | 592
  Race/Ethnicity: Other or Missing | 43 | 33 | 76
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Midwest | 148 | 961 | 1109
  United States: Northeast | 269 | 0 | 269
  United States: Northwest | 274 | 0 | 274
  United States: Southeast | 205 | 339 | 544
Emergency department visits year prior to study [Mean (Standard Deviation); unit: visits] | 1.1 (1.9) | 0.9 (1.7) | 1.0 (1.8)
Inpatient stays year prior to study [Mean (Standard Deviation); unit: stays] | 0.8 (1.6) | 0.4 (1.1) | 0.6 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Any Hospitalization or Any Emergency Room Visits
Description: 24-month count hospitalization and emergency room visits compared between the intervention and usual care groups
Time Frame: 24-months
Measure: Count of Participants; unit: Participants
Groups:
- Control Arm: No intervention. Patients received standard usual care, which generally included the following: nurse coordinators or midlevel practitioners were responsible for general solid organ transplantation (SOT) patient oversight, including ensuring laboratory assessments were scheduled/reviewed and medication regimens were accurate and up to date. For usual care, pharmacists typically were consultants and were only involved in direct patient care if an issue arose, and the nurse or provider engaged the pharmacist for assistance. Within usual follow-up care, pharmacists did not conduct routine daily surveillance of SOT patients.
- Intervention Arm: Patients received the technology-enabled pharmacist intervention in addition to the usual standard of care. The intervention consisted of increased review of patients by a pharmacist and increased scrutiny of patients' medication regimens and laboratory values using a dashboard surveillance system.
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 896 | 1300
Participants
  Any ED Visit During Study | 497 | 574
  Any Inpatient stay During Study | 380 | 391
Statistical Analysis 1: Comparison: Control Arm vs Intervention Arm; Rate of inpatient hospitalization during study; Test type: Superiority; p < .001, Chi-squared
Statistical Analysis 2: Comparison: Control Arm vs Intervention Arm; Test type: Superiority; p < .0001, Chi-squared

2. Secondary Outcome: Total Estimated Health Care Costs, Compared Between the Intervention and Control Groups
Description: 27-month total estimated health care costs, compared between the intervention and control groups (non-zero cost).
  Inpatient cost, outpatient cost, pharmacy cost, total cost
  Time Period (start to censor date) March 01, 2019 to June 30, 2021.
Time Frame: 27-months
Population: The number analyzed in some of the rows of the outcome measure data table differ from the overall number of participants analyzed because not every patient had every type of cost - some didn't have any emergency department (ED) visits, some didn't have any hospitalizations, and a few didn't have any outpatient visits - no visit, no cost.
Measure: Median (Inter-Quartile Range); unit: dollars
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 742 | 1073
dollars
  Inpatient costs: number analyzed (Participants) | 338 | 352
  Inpatient costs | 37,505 [16,797 to 81,891] | 56,600 [22,417 to 108,634]
  Outpatient costs: number analyzed (Participants) | 740 | 1065
  Outpatient costs | 17,077 [6,473 to 38,164] | 25,560 [10,388 to 51,971]
  Pharmacy costs | 10,306 [4,534 to 19,869] | 10,555 [5,374 to 20,485]
  Total costs | 36,255 [15,672 to 80,508] | 51,811 [21,967 to 133,045]
Statistical Analysis 1: Comparison: Control Arm vs Intervention Arm; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Statistical analysis applies to all rows

3. Secondary Outcome: Number of Participants With Graft Survival
Description: Estimated graft survival rates, compared between the intervention and usual care groups and defined as the proportion of patients that continue to have a functioning allograft at the end of the 27-month study
Time Frame: 27-months
Population: All participants who were assigned to the arm
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 896 | 1300
Participants | 864 | 1255
Statistical Analysis 1: Comparison: Control Arm vs Intervention Arm; Test type: Superiority; p = 0.9064, Chi-squared

4. Secondary Outcome: Patient Survival- Percentage of Patients That Died During Study
Description: Estimated patient survival rates, compared between the intervention and usual care groups and defined as the proportion of patients alive at the end of the 27-month study. Number of patients who died during the study (March 2019 - June 2021), Scientific Registry of Transplant Recipients (SRTR) or VA reported.
Time Frame: 27-months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 896 | 1300
Participants | 144 | 195
Statistical Analysis 1: Comparison: Control Arm vs Intervention Arm; Test type: Superiority; p = 0.51, Chi-squared

5. Secondary Outcome: Medication Safety Issues
Description: 23-months, (August 2019-June 2021)
  Potential medication safety issues, defined as the proportion of patients with the following, based on automated reports for the transplant medication dashboard:
  1. Percent of patients with missing labs
  2. Percent of patients alarming lab values without follow up scheduled
  3. Immunosuppression adherence, estimated using the proportion of days covered (PDC)
  4. Percent of patients on significant drug interaction without a immunosuppressant level
  5. Percent of patients with hospital discharge or ED visit without follow up scheduled
Time Frame: 23-months
Population: The dashboard intervention was not utilized in the control group and therefore could not be analyzed for this measure. The number of participants reported in here is inconsistent with total number of participants reported in this arm because there are two levels of analysis, the patient level and at the transplant level. Some patients had multiple transplants. Also, not every patient triggered an alert in the dashboard, so the alert numbers may differ from the number of clinical participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 1,197
Participants
  Percent of patient with missing labs | 733
  Percent of patients alarming lab values without follow up scheduled | 760
  Immunosuppression adherence, estimated using the proportion of days covered (PDC) <80% | 756
  Percent of patients with hospital discharge or ED visit without follow up scheduled | 196

6. Secondary Outcome: Clinically Relevant Alerts
Description: Proportion of alerts that were deemed clinical relevant and actionable by the intervention pharmacists
  22 months (August 2019-June 2021)
Time Frame: 22-months
Population: as for outcome 5
Measure: Count of Units; unit: Dashboard alerts
Units Other Than Participants: Dashboard alerts
Arm/Group | Intervention Arm
Number analyzed (Participants) | 1197
Number analyzed (Dashboard alerts) | 18132
Dashboard alerts | 15013

7. Secondary Outcome: Dashboard-Accepted Interventions
Description: Proportion of interventions that were deemed to be accepted when made to other providers based on dashboard reporting information
  Percentage of patients that had an alert accepted and addressed by a clinician
  23 months, August 2019 - June 2021
Time Frame: 23-months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 1197
Participants
  Patients with an alert that led to a pharmacist conducting a medication change | 102
  Patients with an alert addressed by a non-pharmacist | 570

8. Secondary Outcome: Average Time Responding to Dashboard Alerts
Description: Average time each intervention pharmacist spent on assessing the dashboard alerts per week over the course of 23 months.
Time Frame: 23-months
Population: The dashboard intervention was not utilized in the control group and therefore could not be analyzed for this measure.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Participating Pharmacists in Intervention Arm: Participating pharmacists randomizing into the Intervention arms of the study
Arm/Group | Participating Pharmacists in Intervention Arm
Number analyzed (Participants) | 8
Minutes | 70 (188)

ADVERSE EVENTS:
Time Frame: 27-month study period
Description: Only death and serious adverse events (SAEs) were assessed. SAEs are defined as patients who had an inpatient stay or graft lost during the study.
Groups:
- Control Arm: Usual Care, no intervention.
  The control arm received usual care. Usual care for veteran organ transplant recipients across the 10 study sites is not standardized but generally includes the following: at most sites, nurse coordinators and/ or midlevel practitioners are responsible for general transplant patient oversight, including ensuring laboratory assessments are scheduled/reviewed and medication regimens are accurate and up to date. However, large patient numbers and workload constraints preclude these health care professionals from prospective detailed daily monitoring of patients. Within usual follow-up care, pharmacists do not conduct routine daily surveillance of all transplant patients
Arm/Group | Control Arm | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 144/896 | 195/1300
Serious Adverse Events (participants affected / at risk) | 412/896 | 436/1300
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Arm (N=896) | Intervention Arm (N=1300)
Graft Failure (General disorders) | 32 | 45 — Graft failure during study
Inpatient hospitalization (General disorders) | 380 | 391 — Inpatient stays during study

LIMITATIONS AND CAVEATS:
This was a pragmatic study, utilization of the system was not required and not uniform across sites or pharmacists. Not all alerts produced were addressed or deemed clinically relevant by intervention site pharmacists. Only ED visits and hospitalizations that occurred within the VA system were captured and used for outcome assessment for this study, which is a limitation. SRTR data for acute rejections are not comprehensive as patients were, on average, 9-years post-transplant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT03860818/Prot_SAP_000.pdf